CLINICAL TRIAL: NCT01228747
Title: A Double-blind, Multicenter, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of Adjunctive Treatment With Oral Levetiracetam, in Epilepsy Patients Aged ≥16 Years, With Generalized Tonic-clonic (GTC) Seizures
Brief Title: A Double-blind, Placebo-controlled Study of Levetiracetam in Epilepsy Patients With Generalized Tonic-clonic Seizures (Except Partial Seizures Evolving to Secondarily Generalized Seizures)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N01159; 2014-004401-32 (EudraCT Number)
Record Dates: First submitted 2010-10-22; First posted 2010-10-26 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy; Generalized Tonic-Clonic Seizures
Keywords: Levetiracetam; epilepsy; generalized tonic-clonic
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo for 28 weeks
  Interventions: Drug: Placebo
- Levetiracetam (Experimental): Levetiracetam treatment with flexible dosing of 1000 mg/day or 2000 mg/day or 3000 mg/day for 28 weeks
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Oral dose at flexible increase doses: 1000 mg/day or 2000 mg/day or 3000 mg/day, twice daily, 28 weeks
  Other Names: Keppra®
  Arms: Levetiracetam
Drug: Placebo — Matching oral placebo tablets twice daily for 28 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of levetiracetam treatment used as adjunctive therapy in Japanese and Chinese epilepsy patients aged ≥16 years and with uncontrolled Generalized Tonic-Clonic seizures despite treatment with 1 or 2 anti-epileptic drugs.

ELIGIBILITY:
Inclusion Criteria:

* An epilepsy patient with generalized tonic-clonic seizures that are classifiable according to the ILAE classification of epileptic seizures (Epilepsia, 1981)
* A patient on a stable dose of 1 or 2 anti-epileptic drugs for the last 4 weeks (potassium bromide and sodium bromide for the last 12 weeks) prior to and during the combined baseline period

Exclusion Criteria:

* Presence of any sign (clinical or imaging procedures) suggesting a progressive brain lesion/disease, in particular, progressive disorder with epileptic seizures
* Diagnosis of Lennox-Gastaut Syndrome
* Confirmed focal epilepsy based on clinical signs (seizure types), with consistent electroencephalogram and magnetic resonance imagining features
* A history of convulsive or non-convulsive status epilepticus while taking concomitant anti-epileptic drugs for the last 3 months prior to Visit 1

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2010-10; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (58):
- China (19):
  - 1, Beijing
  - 9, Beijing
  - 12, Changchun
  - 19, Chengdu
  - 6, Chengdu
  - 10, Chongqing
  - 16, Guangzhou
  - 5, Guangzhou
  - 18, Harbin
  - 13, Kunming
  - 22, Nanjing
  - 14, Qingdao
  - 2, Shanghai
  - 3, Shanghai
  - 17, Shenyang
  - 15, Taiyuan
  - 8, Wuhan
  - 20, Xi'an
  - 7, Xi'an
- Japan (39):
  - 152, Fujisawa
  - 112, Fukuoka
  - 113, Fukuoka
  - 166, Fukuoka
  - 187, Fukushima
  - 124, Hamamatsu
  - 175, Higashiosaka
  - 162, Himeji
  - 110, Hiroshima
  - 177, Hiroshima
  - 165, Iizuka
  - 143, Kagoshima
  - 156, Kagoshima
  - 176, Kameda
  - 150, Kashihara
  - 153, Kashiwakazi
  - 105, Kokubunji
  - 172, Miyakonojō
  - 179, Miyazaki
  - 186, Miyazaki
  - 189, Nagoya
  - 106, Niigata
  - 158, Okayama
  - 157, Osaka
  - 174, Osaka
  - 130, Otaru
  - 129, Ōsaka-sayama
  - 170, Saito
  - 147, Sakai
  - 194, Sakai
  - 117, Sapporo
  - 131, Sapporo
  - 304, Sapporo
  - 103, Sendai
  - 168, Shimajiri
  - 138, Shimotsuke
  - 121, Shizuoka
  - 120, Tokyo
  - 111, Ube

REFERENCES:
- [Result] Wu L, Yagi K, Hong Z, Liao W, Wang X, Zhou D, Inoue Y, Ohtsuka Y, Sasagawa M, Terada K, Du X, Muramoto Y, Sano T. Adjunctive levetiracetam in the treatment of Chinese and Japanese adults with generalized tonic-clonic seizures: A double-blind, randomized, placebo-controlled trial. Epilepsia Open. 2018 Sep 29;3(4):474-484. doi: 10.1002/epi4.12255. eCollection 2018 Dec. PMID 30525116
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in Japan and China in October 2010.
Pre-assignment Details: Participant Flow refers to the Randomized Set consisting of all screened subjects who signed the Informed Consent form, participated in the prospective Baseline Period and were randomized at Visit 2.
Groups:
- Levetiracetam: Levetiracetam treatment with dosing of 1000 mg/day or 2000 mg/day or 3000 mg/day for 28 weeks
  Levetiracetam: Oral dose tablets, twice daily
Period: Overall Study
Arm/Group | Placebo | Levetiracetam
Started | 125 | 126
Completed | 60 | 81
Not Completed | 65 | 45
Not completed — Adverse Event | 8 | 4
Not completed — Lack of Efficacy | 40 | 27
Not completed — Protocol Violation | 6 | 5
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Other Reason | 2 | 5

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS), which is a subset of the Randomized Set and consisted of all subjects who received at least 1 dose of study medication after randomization, either Placebo or Levetiracetam.
Groups:
- Placebo: Matching placebo for 28 weeks
  Placebo: Matching oral placebo tablets twice daily
- Total: Total of all reporting groups
Arm/Group | Placebo | Levetiracetam | Total
Number analyzed (Participants) | 125 | 126 | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 10 | 21
  Between 18 and 65 years | 113 | 115 | 228
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (12.5) | 31.5 (11.3) | 32.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 47 | 96
  Male | 76 | 79 | 155
Region of Enrollment [Number; unit: participants]
  China | 104 | 104 | 208
  Japan | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From the Combined Baseline in the Generalized Tonic-clonic Seizure Frequency Per Week Over the 28-week Treatment Period (Dose Adjustment + Evaluation Periods)
Description: Percentage change in generalized tonic-clonic (GTC) seizure frequency per week from Combined Baseline B over the Treatment Period A is calculated using the equation:
  Percentage change from Baseline = ((A-B)/B)*100. Percentage change from baseline is not defined for subjects whose baseline information is missing / unknown or equal to zero, or whose seizure frequency per week is missing / unknown. A negative value in change in generalized tonic-clonic (GTC) seizure frequency indicates a reduction of generalized tonic-clonic (GTC) seizure frequency over the 28-week treatment Period.
  Combined Baseline means: a 4-week Retrospective Baseline + 4-week Prospective Baseline or 8-week Prospective Baseline
Time Frame: From Baseline to Week 28
Population: Full Analysis Set consisted of all subjects in the SS who had an evaluable Baseline and at least 1 post-Baseline GTC seizure count data point for the primary efficacy analysis excluding those who had seriously violated GCP. Evaluable Baseline for the primary efficacy analysis: at least 1 GTC seizure was documented for the Combined Baseline.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Placebo | Levetiracetam
Number analyzed (Participants) | 109 | 117
Percentage Change | -13.19 (55.54) | -68.22 (34.95)
Statistical Analysis 1: Comparison: Placebo vs Levetiracetam; The statistical hypotheses, null hypothesis (H0) and alternate hypothesis (H1), are stated below: H0: μLEV = μPBO vs. H1: μLEV ≠ μPBO ANCOVA on the endpoint "percentage change from Combined Baseline of GTC seizures per week" using "treatment" and "country" as factors (categorical predictors) and "Combined Baseline GTC seizure frequency per week" as a covariate (a continuous predictor) where μLEV and μPBO are adjusted means for LEV and PBO, respectively; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was 2-sided, and was performed using a significance (α) level of 0.05; Mean Difference (Net) = -56.13, 95% CI 2-sided [-68.24 to -44.02], Standard Error of Mean 6.15

2. Secondary Outcome: The Percentage Change in Generalized Tonic-clonic Seizure Frequency Per Week From the Combined Baseline Over the Evaluation Period
Description: Percentage change in generalized tonic-clonic (GTC) seizure frequency per week from combined baseline B over the Evaluation Period A is calculated using the equation:
  Percentage change from Baseline = ((A-B)/B)*100. Percentage change from baseline is not defined for subjects whose baseline Information is missing / unknown or equal to zero, or whose seizure frequency per week is missing / unknown. A negative value in change in generalized tonic-clonic (GTC) seizure frequency indicates a reduction of generalized tonic-clonic (GTC) seizure frequency.
  Combined Baseline means: a 4-week Retrospective Baseline + 4-week Prospective Baseline or 8-week Prospective Baseline.
Time Frame: From Baseline to Evaluation Period (Week 12 to Week 28)
Population: Of the 226 subjects in the Full Analysis Set (FAS), 205 are included in the analysis of this Outcome Measure in Evaluation Period.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Placebo | Levetiracetam
Number analyzed (Participants) | 97 | 108
Percentage Change | -4.44 (153.82) | -68.27 (42.63)

3. Secondary Outcome: Generalized Tonic-clonic Seizures 50 % Responder Rate (the Proportion of Subjects With 50 % or More Reduction From the Combined Baseline in the Frequency of Generalized Tonic-clonic Seizures) During the Treatment Period
Description: A subject with an at least 50 % reduction in weekly generalized tonic-clonic (GTC) seizure frequency from Combined Baseline Period to the Treatment Period is considered a GTC 50 % responder.
  Combined Baseline means: a 4-week Retrospective Baseline + 4-week Prospective Baseline or 8-week Prospective Baseline
Time Frame: From Baseline to Week 28
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Levetiracetam
Number analyzed (Participants) | 109 | 117
participants | 31 | 91

4. Secondary Outcome: Generalized Tonic-clonic Seizures 50 % Responder Rate (the Proportion of Subjects With 50 % or More Reduction From the Combined Baseline in the Frequency of Generalized Tonic-clonic Seizures) During the Evaluation Period
Description: A subject with an at least 50 % reduction in weekly generalized tonic-clonic (GTC) seizure frequency from Combined Baseline Period to the Evaluation Period is considered a GTC 50 % responder.
  Combined Baseline means: a 4-week Retrospective Baseline + 4-week Prospective Baseline or 8-week Prospective Baseline
Time Frame: From Baseline to Evaluation Period (Week 12 to Week 28)
Population: Of the 226 subjects in the Full Analysis Set (FAS), 205 are included in the analysis of this Outcome Measure.
Measure: Number; unit: participants
Arm/Group | Placebo | Levetiracetam
Number analyzed (Participants) | 97 | 108
participants | 33 | 82

5. Secondary Outcome: Generalized Tonic-clonic Seizure Freedom Over the Evaluation Period
Description: A subject with a non-missing weekly generalized tonic-clonic (GTC) baseline seizure frequency and a weekly GTC seizure frequency of zero throughout the Evaluation Period, is considered as a GTC seizure-free subject on the Evaluation Period.
Time Frame: Evaluation Period (Week 12 to Week 28)
Population: Of the 226 subjects in the Full Analysis Set (FAS), 205 are included in the analysis of this Outcome Measure.
Measure: Number; unit: participants
Arm/Group | Placebo | Levetiracetam
Number analyzed (Participants) | 97 | 108
participants | 3 | 32

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the Prospective Baseline Period ( Week -8 to Week 0) over Dose Adjustment (12 weeks) and Evaluation Period (16 weeks) until Conversion or Withdrawal Period (4-6 weeks).
Description: Adverse Events refer to the Safety Set (SS), which is a subset of the Randomized Set and consisted of all subjects who received at least 1 dose of study medication after randomization, either Placebo or Levetiracetam.
  Adverse Events were presented for the Dose Adjustment and Evaluation Period.
Arm/Group | Placebo | Levetiracetam
Serious Adverse Events (participants affected / at risk) | 4/125 | 1/126
Other Adverse Events (participants affected / at risk) | 32/125 | 40/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=125) | Levetiracetam (N=126)
Drowning (General disorders) | 2 (2) | 0 (0)
Sudden unexplained death in epilepsy (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=125) | Levetiracetam (N=126)
Pyrexia (General disorders) | 5 (5) | 7 (8)
Nasopharyngitis (Infections and infestations) | 20 (36) | 24 (33)
Platelet count decreased (Investigations) | 4 (4) | 7 (8)
Protein urine present (Investigations) | 1 (1) | 10 (11)
Dizziness (Nervous system disorders) | 9 (14) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days